CLINICAL TRIAL: NCT06016244
Title: Safe, Effective and Cost-Effective Oxygen Saturation Targets for Children and Adolescents With Respiratory Distress: a Randomized Controlled Trial
Acronym: OxyKids
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Spaarne Gasthuis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022.0100; 2023-504817-56 (Other: EMA CTIS NR)
Record Dates: First submitted 2023-07-31; First posted 2023-08-29 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-02

CONDITIONS: Bronchiolitis; Lower Respiratory Tract Infection; Bronchial Hyperreactivity
Keywords: Oxygen saturation target; SpO2; Children
MeSH Terms: conditions — Bronchiolitis; Bronchial Hyperreactivity

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial, parallel group, block randomized and stratified by age and centre.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 88% oxygen saturation threshold (Experimental): Patients in this arm will receive supplemental oxygen when SpO2 falls below 88% or when other clinical symptoms indicate a need for supplemental oxygen.
  Interventions: Other: Oxygen saturation threshold
- 92% oxygen saturation threshold (Active Comparator): Patients in this arm will receive supplemental oxygen when SpO2 falls below 92% or when other clinical symptoms indicate a need for supplemental oxygen.
  Interventions: Other: Oxygen saturation threshold

INTERVENTIONS:
Other: Oxygen saturation threshold — Oxygen saturation threshold on which supplemental oxygen is decided

SUMMARY:
The goal of this clinical trial is to find out at which lower limit for saturation (amount of oxygen in the blood) we can best give extra oxygen to children that have been admitted for shortness of breath. We hope to accomplish a shorter period of illness for these children and that they can be discharged home earlier. Participants will receive supplemental oxygen if their blood oxygen levels are below 88% or below 92%. After admission, (parents of) participating children will fill out questionnaires. We will compare the two groups on their hospitalization duration and recovery.

In other words, is it better to maintain a lower limit of 88% saturation or a lower limit of 92% in children admitted for shortness of breath?

ELIGIBILITY:
Inclusion Criteria:

* 6 weeks to 12 years of age (corrected age for children with gestational age < 37 weeks)
* hospitalized with respiratory distress due to bronchiolitis, viral wheeze or lower respiratory tract infection, as diagnosed by the treating physician. Viral wheeze can only be diagnosed below the age of 6 years.
* requiring supplemental oxygen as per usual care (SpO2 <92% or for treating symptoms of respiratory distress as determined by the treating physician

As respiratory distress in children with an asthma attack is mainly driven by hypoxia, they are at risk of undertreatment in the acute phase of the attack. Therefore, children aged 6-12 years of age with an asthma attack are excluded from this study.

Exclusion Criteria:

* children with, except for the studied diseases, pre-existing cardiopulmonary, neurological or hematological conditions (e.g. congenital thoracic malformation, airway malacia, post infectious bronchiolitis obliterans, childhood interstitial lung disease. primary immune deficiency)
* children born <32 weeks gestational age
* children already included in other studies, which potentially interfere with this study
* children (of parents) without a stable internet connection needed for answering questionnaires
* children previously included in the current study
* considering questionnaires are only available in Dutch and English, children (of parents) with different languages will be excluded.

Ages: 6 Weeks to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 560 (Estimated)
Dates: Start 2023-09-04 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to meeting all discharge criteria | Discharge criteria are checked daily during admission up to discharge (generally a few days up to a week but longer if admission lasts longer) and the time and date at which all discharge criteria have been met will be recorded.
  Time in hours from admission to meeting all discharge criteria
  Discharge criteria include:
  * No need for supplemental oxygen for 4 hours, including a period of sleep for children aged < 2 years
  * Clinically fit for discharge with normal or minimally increased respiratory rate AND no or mild respiratory distress, as judged by nurses and physicians using the Parshuram et al scoring system, commonly used in Dutch paediatric practice as part of the Pediatric Early Warning Scale].
  * No need for in-hospital feeding or medication by nasogastric tube (NGT).
  * No need for in-hospital intravenous treatment.
  * No need for in-hospital nebulized bronchodilator treatment.
  * No need for in-hospital treatment with metered dose inhalator inhalations more often than every 3 hours.
  * No need for high flow delivered by high flow nasal cannula or nasal prongs.

SECONDARY OUTCOMES:
Length of stay | During admission
  Time from admission to discharge in hours
Pediatric Intensive Care Unit (PICU) admissions | During admission
  Number of PICU admissions per group
Time on oxygen therapy | During admission
  Time in hours spent on supplemental oxygen
Duration of symptoms | from admission to 90 days after discharge
  Measured as days from admission to having met all of the following criteria: resolution of cough, resolution of dyspnea as indicated by parent, cessation of scheduled bronchodilator use.
Return to normal health | from admission to 90 days after discharge
  Measured as days from admission to parent reported normal health. Upon discharge parents/patients are asked to record the last day of illness and report this in the follow-up questionnaires
Time to return to school/daycare | from admission to 90 days after discharge
  Measured as days from admission to parent reported return to school/daycare
Unscheduled health care visits or admissions after discharge | from admission to 28 days after discharge
  Number of unscheduled visits or admissions up to 28 days after discharge
Patient quality of life | at discharge, 7, 28 and 90 days follow-up
  Measured by digital questionnaire of EQ-5D-Y (modified versions are used in agreement with EuroQol for patients < 4 years)
Overall pediatric health | at discharge, 7, 28 and 90 days follow-up
  ICHOM PROMIS Pediatric Global Health set
Parental anxiety | at discharge, 7 and 28 days follow-up
  by anxiety items of Hospital Anxiety and Depression Scale
Economic evaluation | Up to 90 days after discharge
  The aim of the economic evaluation is to relate the incremental costs of an SpO2 of 88% (intervention) in comparison with an SpO2 of 92% (control) to the incremental health effects. Both a cost-effectiveness analysis (CEA) and a cost-utility analysis (CUA) will be performed from a societal and healthcare perspective

OTHER OUTCOMES:
Skin type influence | Up to 90 days after discharge
  Investigation in to the influence of skin type on safety and effectiveness outcomes
Time spent in 88%-92% window | recorded at discharge based on monitoring data registered during admission, generally a few days to a week but longer if admission lasts longer.
  Time spent in 88%-92% saturation window, measured by extracted continous monitoring data from patients where this is technically a possibility.

CONTACTS AND LOCATIONS:
Overall Officials: Annmeie LM Boehmer, MD, PhD, Principal Investigator — Spaarne Gasthuis
Locations (9):
- Netherlands (9):
  - Spaarne Gasthuis, Haarlem, North Holland
  - Canisius Wilhelmina Ziekenhuis, Arnhem
  - Rijnstate Ziekenhuis, Arnhem
  - Amphia Ziekenhuis, Breda
  - Martini Ziekenhuis, Groningen
  - Tergooi Ziekenhuis, Hilversum
  - St Antonius Ziekenhuis, Nieuwegein
  - Franciscus Gasthuis en Vlietland, Rotterdam
  - Isala Klinieken, Zwolle

IPD SHARING:
Plan to Share IPD: Yes
Data and metadata will be made available for reuse after removing data from participants who did not consent to reuse of their data and removing any potentially identifiable data. Data archiving and sharing will be done through DANS EASY. The Dublin Core metadata scheme will be used.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: The data will only be made available for reuse after completion of the study and all planned publications of the results.
Access Criteria: Other researchers will be able to find the metadata in the data repository. They could express their interest in the dataset through emailing the PI. After meeting the sharing and reuse conditions and approval of the PI, data access will be provided through the data repository.

REFERENCES:
- [Derived] Louman S, van Stralen KJ, Koppelman G, Vaessen-Verberne A, Bekhof J, Bosmans J, Brackel C, Kamps AWA, de Kleer I, Balemans W, Scheffer M, Brouwer M, van den Beukel M, Andrinopoulou ER, Pijnenburg MWH, Boehmer ALM. Safe, effective and cost-effective oxygen saturation targets for children and adolescents with respiratory distress: protocol for a randomised controlled trial (OxyKids study). BMJ Open. 2024 Dec 22;14(12):e087891. doi: 10.1136/bmjopen-2024-087891. PMID 39806594